CLINICAL TRIAL: NCT05157230
Title: Evaluation of Deltoid Muscle Exercises on Injection Site and Arm Pain After Pfizer - BioNTech (BNT162b2) COVID - 19 Vaccination, A Randomized Controlled Study
Brief Title: Evaluation of Deltoid Exercises on Injection Site Pain After (BNT162b2) COVID - 19 Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zulfı engındenız, Zulfi Engindeniz, MD, Principal investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-KAEK-25 2021/08-21
Record Dates: First submitted 2021-12-11; First posted 2021-12-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Vaccines, Adverse Effects; Injection Site Reaction
Keywords: BNT162B2; exercise; Injection Site Reaction; Pain Management
MeSH Terms: conditions — Injection Site Reaction; Motor Activity; Agnosia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): volunteers in this group do shoulder/arm exercises after vaccine injection and fill in the pain diary
  Interventions: Behavioral: exercise
- no-exercise (No Intervention): volunteers in this arm only completed the pain diary without any intervention

INTERVENTIONS:
Behavioral: exercise — volunteers in the exercise arm instructed to do three basic deltoid muscle exercises 3 times daily at least 20 repetitions for each exercise for five days. exercises were side lateral shoulder raises, front shoulder raises with hyperextension and mid range arm circles.
  Arms: exercise

SUMMARY:
Pfizer - BioNTech (BNT162b2) COVID - 19 vaccine is the first vaccine to be approved for emergency use by FDA. The most commonly reported side effect of the BNT162b2 vaccination is mild-to-moderate pain at injection site, i.e. deltoid muscle. Injection site pain may be observed during and after vaccine injection, and severity of pain may vary according to the type of vaccine, patients age, sex, level of anxiety, needle size, injection site and technique and patient positioning. Vaccination pain is one of the reasons of vaccine hesitancy and World Health Organization (WHO) recommended various measures to mitigate pain at the time of vaccination.

Exercise is one of the suggested methods to relieve the pain and anxiety in various conditions including vaccination site pain. However, we found no studies addressing injection site pain after the vaccination and pain associated with BNT162b2 vaccine. Aim of our study is to evaluate effectiveness of deltoid muscle exercises to relieve injection site pain observed after BNT162b2 vaccination.

DETAILED DESCRIPTION:
The study was started at the designated COVID - 19 vaccination department of Bursa Yuksek Ihtisas research and training hospital Approvals was obtained from Republic of Turkey Ministry of Health and institutional review board and ethics committee and the study was conducted in concordance with Declaration of Helsinki.

Volunteers were selected among the healthy persons who admitted to our vaccination department to have BNT162b2 vaccine. Selection criteria were age being over 18, having no physical disability to perform the physical exercises given and willingness to participate in the study and sign an informed consent. People under the age of 18, patients with conditions that prevent them doing the exercises given and who did not want to participate in the study were excluded from the study.

Volunteers who accept to participate in the study, were randomized in to exercise vs. no-exercise groups according to a previously formed online randomization list. All volunteer's demographic data and vaccination status (first or second dose) were recorded. Both groups were asked to keep a five - day pain diary using numeric rating scale (NRS) and to also record any use of analgesics, any hospital admissions, any side effects other than injection site and arm pain and the time of cessation of pain.

ELIGIBILITY:
Inclusion Criteria:

* vaccination with Bnt162b2
* having no physical disability to perform the physical exercises given
* willingness to participate in the study and sign the informed consent form

Exclusion Criteria:

* vaccination with vaccines other than Bnt162b2
* having physical disability to perform the physical exercises given
* not willing to participate in the study and sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
time to no pain at injection site or arm | within 5 days after vaccination
  time frame between the time of vaccination and self reported time of being pain free

SECONDARY OUTCOMES:
use of analgesics | within 5 days after vaccination
  self reported use of any analgesics
hospital admission | within 5 days after vaccination
  self reported admission to hospital for reasons related to vaccination
mean daily pain score | within 5 days after vaccination
  difference in mean daily pain score in numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Zulfi Engindeniz, MD, Principal Investigator — Bursa Yuksek Ihtisas Reseach and Training Hospital
Locations (1):
- BursaYuksek Ihtisas Research and Training Hospital, Bursa, Turkey (Türkiye)